CLINICAL TRIAL: NCT02016443
Title: Investigation of the Effectiveness of Tizanidine on Pain After Herniorrhaphy
Brief Title: Tizanidine and Pain After Herniorrhaphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIZANIDINE
Record Dates: First submitted 2013-10-10; First posted 2013-12-20 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2013-10

CONDITIONS: Unilateral Inguinal Hernia
Keywords: inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — tizanidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tizanidine (Experimental): Group Tizanidine (Group T) will receive 4 mg tizanidine per oral twice a day during the postoperative first week and the first dose will be administered 1 hour before surgery
  Interventions: Drug: Tizanidine
- Placebo (Placebo Comparator): Group Placebo (Group P) will receive placebo per oral twice a day during the postoperative first week and the first dose will be administered 1 hour before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tizanidine — Group Tizanidine (Group T) will receive 4 mg tizanidine per oral twice a day during the postoperative first week and the first dose will be administered 1 hour before surgery
  Other Names: Sirdalud
  Arms: Tizanidine
Drug: Placebo — Group Placebo (Group P) will receive a placebo per oral twice a day during the postoperative first week and the first dose will be administered 1 hour before surgery
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
Herniorrhaphy is the most frequent general surgical procedure. There are moderate pain complaints after herniorrhaphy. Besides causing discomfort to the patients, pain, can delay recovery and discharge and cause cognitive dysfunction and difficulty with returning to normal daily activity.

A combination of analgesics with different effect sites can reduce the doses needed and analgesic related side effects which is called multimodal analgesia .

Opioids, acetaminophen, nonsteroid anti-inflammatory drugs and cox-2 inhibitors, alfa-2 receptor agonists, steroids, gabapentin and pregabalin have been used for this purpose(4).

Tizanidine is an alfa-2 receptor agonist, and is used for musculoskeletal pain conditions. Tizanidine reduced the local anesthetic requirement in spinal anesthesia.

The aim of this study is to investigate the hypothesis that: Tizanidine can reduce the pain scores, analgesic consumption, analgesic related side effects and provide early return to normal daily activity compared to placebo after inguinal herniorrhaphy.

DETAILED DESCRIPTION:
Age, body mass index (BMI), concomitant diseases, and the ASA physiologic state will be recorded.

Simple randomization will be accomplished with a computer-generated sequence of numbers and sealed envelopes will be used to allocate patients into 2 groups.

Patients in GroupTizanidine will receive 4 mg tizanidine per oral twice a day during the postoperative first week and the first dose will be administered 1 hour before surgery, patients in Group Placebo will receive the same treatment with a placebo pill concurrently with a standard analgesic treatment: dexketoprofen trometamol; 25 mg intravenous (iv) before the induction of anesthesia and 25 mg per oral 3 times a day-1 week and acetaminophen; 1 g iv at the end of surgery. All patients will be instructed to use acetaminophen 500 mg up to 4 times a day for rescue analgesia and to contact the hospital if they have pain despite all three medications.

Heart rate (HR), peripheral oxygen saturation (SpO2), systolic arterial pressure (SAP), diastolic arterial pressure (DAP) and mean arterial pressure (MAP), end tidal CO2 pressure (EtCO2). Baseline values will recorded.

Anesthesia induction and muscle relaxation will be standardized with 2 mg kg-1 propofol, 0.6 mg kg-1 rocuronium and 50 µg fentanyl. Anesthesia will be maintained with oxygen in nitrous oxide and desflurane. The desflurane concentration will be titrated to keep BIS between 40-60. The patients will receive 50 µg fentanyl boluses in case hemodynamic variables changed ≥30% from baseline values. Hypotension will be defined as ≥20% decrease in MAP from baseline values and will be treated with fluid boluses and/or ephedrine. Bradycardia will be defined as a heart rate <50 beat min and will be treated with atropine. All treatments will be recorded. At the end of surgery volatile anesthesia will be discontinued and the patients will be extubated according to clinical extubation criteria. The time elapsed from discontinuation of volatile anesthesia to eye opening with verbal commands will be recorded as time to emergence. The patients will be transferred to the post anesthesia care unit (PACU). The modified Aldrete score will be used to evaluate recovery in the PACU and the patients will be discharged from the PACU when the Aldrete score is ≥9 ( ). Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 1, 6, 12 and 24 hours postoperatively.

During the control visit 1 week after surgery total analgesic consumption and analgesic related adverse events (nausea, vomiting, dizziness…) will be evaluated. Difficulty with normal daily activity will also be evaluated during this visit with the Likert score (1. no difficulty, 2. mild difficulty, 3. difficulty, 4. severe difficulty, 5. unable to perform daily activity due to pain). Health related quality of life will also be evaluated 1 month after surgery; the Short Form (SF)-36 will be used for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing unilateral inguinal herniorrhaphy

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* recurrent hernias
* emergency cases

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 1, 6 and 24 hours postoperatively.
Visual analog pain score | postoperative 6th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 1, 6 and 24 hours postoperatively.
Visual analog pain score | Postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 1, 6 and 24 hours postoperatively.
Visual analog pain score | Postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 1, 6 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Likert score | Postoperative 1 week
  Difficulty with normal daily activity will be evaluated during the first week control visit with the Likert score (1; no difficulty, 2; mild difficulty, 3; difficulty, 4; severe difficulty, 5; unable to perform daily activity due to pain
SF-36 score | Postoperative first month
  Health related quality of life will be evaluated 6 weeks after surgery; the SF-36 will be used for this purpose

OTHER OUTCOMES:
hemodynamic parameters | intraoperative with 5 minutes intervals
  systolic, diastolic, mean arterial pressures and heart rate will be measured with 5 minutes intervals
total analgesic consumption | postoperative 1 week
  total analgesic consumption will be determined at postoperative 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazicioglu, Dr, Principal Investigator — Ministry of Health
Locations (1):
- Diskapi Yildirim Beyazit training and research hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Ward A, Brenner M. Guanylate cyclase from Dictyostelium discoideum. Life Sci. 1977 Oct 1;21(7):997-1008. doi: 10.1016/0024-3205(77)90267-3. No abstract available. PMID 22014
- [Background] Roseboom H, Perrin JH. Oxidation kinetics of phenothiazine and 10-methylphenothiazine in acidic medium. J Pharm Sci. 1977 Oct;66(10):1392-5. doi: 10.1002/jps.2600661010. PMID 21948
- [Derived] Yazicioglu D, Caparlar C, Akkaya T, Mercan U, Kulacoglu H. Tizanidine for the management of acute postoperative pain after inguinal hernia repair: A placebo-controlled double-blind trial. Eur J Anaesthesiol. 2016 Mar;33(3):215-22. doi: 10.1097/EJA.0000000000000371. PMID 26555871